CLINICAL TRIAL: NCT02904733
Title: Validation Study of mHealth Technology in HIV to Improve Empowerment and Healthcare Utilisation: Research and Innovation to Generate Evidence for Personalised Care (EmERGE)
Acronym: EMERGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Brighton and Sussex University Hospitals NHS Trust (Other); Instituut Voor Tropische Geneeskunde (ITM), Antwerp, Belgium. (Unknown); Klinika za infektivne bolesti (KIB), Zagreb, Croatia (Unknown); Centro Hospitalar de Lisboa Central (Other); Fundacion Clinic per a la Recerca Biomédica (Other); University of Brighton (Other); Podmedics, ( POD), Northwood, United Kingdom (Unknown); Universidad Politecnica de Madrid (Other); National Prospective Monitoring System HIV Health-economics Collaboration, (NPMS), Richmond, United Kingdom (Unknown); European Aids Treatment Group (EATG), Brussels, Belgium (Unknown); mHealth Futures LTD, Brighton, United Kingdom (Unknown)
Responsible Party: Principal Investigator, Agathe LEON, Dr, Fundacion Clinic per a la Recerca Biomédica
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: EMERGE
Record Dates: First submitted 2016-07-07; First posted 2016-09-19 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mHealth platform (Experimental): Stable HIV-1 infected subjects will be followed-up using an mHealth platform. The platform will provide users with web based and mobile device applications which interface securely with relevant medical data and facilitate remote access to healthcare providers. The minimum length of follow-up will be 12 months and the maximum 35 months.
  Interventions: Other: mHealth platform

INTERVENTIONS:
Other: mHealth platform — Use of a mHealth platform to inform and empower patient of hies/her own health

SUMMARY:
A large (3900 patients) cohort study, undertaken in five European sites to validate in a mHealth platform to enable self-management of HIV in patients with stable disease using a tailored HTA process, Model for Assessment of Telemedicine Applications (MAST), specifically developed for the assessment of mHealth solutions.

As site recruitment will be sequential and the recruitment period will last 18 months, a maximum follow-up of 35 Months will be undertaken. Study visits will take place at baseline defined as the time of mHealth introduction, months 6, 12, 18, 24 and 30.

DETAILED DESCRIPTION:
Number of Study Centres: 5 Duration of Study: 35 Months Criteria for Evaluation: Usability of the mHealth platform, patient self-management and empowerment, clinical safety (virological suppression maintenance, CD4 count, laboratory parameters, adverse events and adherence), quality of life and self-economy will be assessed by questionnaires and laboratory parameters.

Routine data on patient demographics, treatment and investigations which will include viral load, CD4, haematology, biochemistry and urine sample. Patient Activation Measure, Quality of life, adherence questionnaire and economic questionnaires will be performed at baseline and at months 12 and 24. Satisfaction System Usability Scale will be evaluated at month 12 and 24.

ELIGIBILITY:
Inclusion Criteria:

1. Documented HIV-1 infection
2. Aged at least 18 years old
3. Able to give informed consent
4. In possession of a smartphone, tablet, or similar technology supporting the mHealth platform
5. Stable on ART: Defined as ART should be unchanged for at least 3 months and viral load undetectable (<50 copies/ml) for at least 6 months.
6. Clinically stable from an HIV perspective: Defined as without opportunistic infection or AIDS related cancers within the previous 12 months

Exclusion Criteria:

1. Aged less than 18 years
2. Pregnant
3. Participating in a clinical trial or receiving an investigational medication
4. Unable to comprehend the patient information sheet
5. Unable to comprehend the instructions for using the mHealth platform
6. Considered for any other reason by their regular physician to be unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3900 (Estimated)
Dates: Start 2017-04-07 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Changes in Patient Activation Measure (PAM-13) questionnaire from baseline | months 12 and 24

SECONDARY OUTCOMES:
Changes in Satisfaction System Usability Scale (SUS) | months 12 and 24
Maintenance of virological suppression (HIV-1 RNA <50 c/ml) | months 12 and 24
Change in CD4 count | months 12 and 24
Change in blood lipid profile | months 12 and 24
Changes in Quality of life (EQ-5D-5L questionnaire) from baseline | months 12 and 24
Changes in Quality of life (PROQOL-HIV questionnaire) from baseline | months 12 and 24
Changes in adherence quantified by Morisky-Green questionnaire | months 12 and 24
Percentage of patients with changes in ART from baseline | months 12 and 24
Changes on self-reported economic questionnaire aspects from baseline | months 12 and 24

CONTACTS AND LOCATIONS:
Locations (5):
- Prins Leopold Instituut Voor Tropische Geneeskunde, Antwerp, Belgium
- Klinika za Infektivne Bolesti Dr. Fran Mihaljevic, Zagreb, Croatia
- Centro Hospitalar de Lisboa Central, Lisbon, Portugal
- Hospital Clínic i Provincial, Barcelona, Spain
- University of Brighton, Brighton, United Kingdom